CLINICAL TRIAL: NCT07301255
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, 12-Week Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of ENV-294 in Adult Participants With Moderate-to-Severe Asthma
Brief Title: ENV-294 for Moderate-to-Severe Asthma: A 12-Week Study in Adults
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Enveda Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ENV-294-211
Record Dates: First submitted 2025-12-10; First posted 2025-12-24 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Asthma
Keywords: Asthma in Adults
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ENV-294 Treatment Arm (Experimental): Participants will be treated with ENV-294 if they are randomized to this treatment arm.
  Interventions: Drug: ENV-294
- Placebo Arm (Placebo Comparator): Participants will be treated with placebo (matching the appearance of ENV-294 active drug) if they are randomized to the placebo arm.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ENV-294 — ENV-294 is an orally administered investigational capsule formulation. Participants receive 800 milligrams (mg) once daily by mouth for 12 weeks. Capsules are taken with water, at approximately the same time each day, with or without food.
  Arms: ENV-294 Treatment Arm
Drug: Placebo — Matching oral capsule that does not contain active drug. Administered once daily by mouth for 12 weeks under the same conditions as the investigational product.
  Arms: Placebo Arm

SUMMARY:
This study will evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and potential efficacy of ENV-294 in adults with moderate to severe asthma who are receiving background treatment with inhaled corticosteroids (ICS) and long-acting beta₂-agonists (LABA).

Participants will take oral ENV-294 or placebo once daily for 12 weeks. The study includes a screening period of up to 28 days before randomization to confirm eligibility. Study visits and assessments will be conducted to monitor safety, measure drug levels in the blood, and evaluate effects on asthma control and lung function.

ELIGIBILITY:
Inclusion Criteria:

* Able to read, understand, and sign an informed consent form before any study procedures.
* Male or female adults aged 18 to 75 years with a physician diagnosis of moderate to severe asthma for at least 12 months.
* Receiving stable treatment with an inhaled corticosteroid (ICS) plus a long-acting beta₂-agonist (LABA) for at least 2 months before screening.
* Pre-bronchodilator FEV₁ between 50% and 80% of predicted normal at screening and baseline.
* Demonstrated bronchodilator reversibility, defined as ≥12% and ≥200 mL improvement in FEV₁ (or ≥20% increase in peak expiratory flow) after short-acting bronchodilator use.
* ACQ-5 score ≥1.25 and ≤3.0 at screening and baseline.
* History of at least one asthma exacerbation in the past 12 months requiring systemic corticosteroids or hospitalization/emergency care.

Exclusion Criteria:

* Had a moderate or severe asthma exacerbation within 4 weeks before screening.
* Have a history of life-threatening asthma, including intubation or respiratory arrest.
* Have any other significant pulmonary disease (e.g., COPD, bronchiectasis, pulmonary fibrosis, cystic fibrosis, tuberculosis, lung cancer, or eosinophilic syndromes).
* Had bronchial thermoplasty within 2 years before screening.
* Used biologic therapies for asthma (e.g., benralizumab, mepolizumab, reslizumab, omalizumab, dupilumab, or tezepelumab) within 6 months or 5 half-lives prior to baseline.
* Require immunosuppressive medications or frequent systemic corticosteroids (more than 3 courses in the past 6 months).
* Are current smokers or former smokers with >10 pack-year history or who quit within 6 months before screening.
* Have uncontrolled hypertension (systolic ≥160 mmHg or diastolic >95 mmHg).
* Have significant hepatic impairment or any other condition that, in the investigator's opinion, would interfere with study participation or interpretation of results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Incidence and Severity of Adverse Events | From first dose through approximately 16 weeks
  Number and percentage of participants with treatment-emergent adverse events (AEs), serious adverse events (SAEs), and adverse events leading to discontinuation of study drug. Events will be summarized by severity and relationship to study treatment.
Change from baseline in hemaglobin. | Baseline through approximately 16 weeks (end of study).
  Assessment of change from baseline in hemoglobin concentration to evaluate the safety and tolerability of ENV-294.
Observed values, change from baseline, and percent change from baseline in heart rate (beats per minute) as a measure of safety and tolerability of ENV-294. | Baseline through approximately 16 weeks (end of study).
  Heart rate measured from 12-lead ECG recordings in beats per minute to assess cardiac safety and tolerability.
Observed value, change from baseline, and percent change from baseline in systolic blood pressure (mmHg) as a measure of safety and tolerability. | Baseline through approximately 16 weeks (end of study).
  Systolic blood pressure measured in millimeters of mercury (mmHg) using standard clinical procedures at each study visit to assess safety and tolerability of ENV-294.
Change from baseline in clinical chemistry laboratory values | Baseline through approximately 16 weeks (end of study).
  Evaluation of changes from baseline in serum clinical chemistry values - including electrolytes (sodium, potassium, chloride), liver function tests (ALT, AST, alkaline phosphatase, bilirubin), kidney function tests (creatinine, blood urea nitrogen), and glucose - to assess the safety and tolerability of ENV-294.
Observed values and change from baseline in coagulation parameters as primary measures of safety and tolerability of ENV-294. | Baseline through approximately 16 weeks (end of study).
  Coagulation tests include prothrombin time (PT), activated partial thromboplastin time (aPTT), and international normalized ratio (INR). Changes from baseline will be assessed to evaluate safety and tolerability of ENV-294.
Observed values and change from baseline in urinalysis parameters as primary measures of safety and tolerability of ENV-294. | Baseline through approximately 16 weeks (end of study).
  Urinalysis parameters include color, clarity, specific gravity, pH, protein, glucose, ketones, blood, leukocytes, and microscopic evaluation, as applicable. Changes from baseline will be evaluated to assess safety and tolerability of ENV-294.
Observed values, change from baseline, and percent change from baseline in RR interval (milliseconds) as a measure of safety and tolerability of ENV-294. | Baseline through treatment and end of study (approximately Week 16).
  RR interval measured from 12-lead ECGs in milliseconds (ms) to assess cardiac safety and tolerability.
Observed values, change from baseline, and percent change from baseline in PR interval (milliseconds) as a measure of safety and tolerability of ENV-294. | Baseline through treatment and end of study (approximately Week 16).
  PR interval measured in milliseconds (ms) using standard 12-lead ECGs to assess safety and tolerability.
Observed values, change from baseline, and percent change from baseline in QRS duration (milliseconds) as a measure of safety and tolerability of ENV-294. | Baseline through treatment and end of study (approximately Week 16).
  QRS duration measured in milliseconds (ms) using standard 12-lead ECGs to assess cardiac conduction and safety.
Observed values, change from baseline, and percent change from baseline in QT interval (milliseconds) as a measure of safety and tolerability of ENV-294. | Baseline through treatment and end of study (approximately Week 16).
  QT interval measured in milliseconds (ms) using standard 12-lead ECGs to assess cardiac repolarization safety.
Observed values, change from baseline, and percent change from baseline in QTc Bazett (milliseconds) as a measure of safety and tolerability of ENV-294. | Baseline through treatment and end of study (approximately Week 16).
  QTc Bazett (QT corrected for heart rate using Bazett's formula) measured in milliseconds (ms) to evaluate cardiac safety.
Observed values, change from baseline, and percent change from baseline in QTc Fridericia (milliseconds) as a measure of safety and tolerability of ENV-294. | Baseline through treatment and end of study (approximately Week 16).
  QTc Fridericia (QT corrected for heart rate using Fridericia's formula) measured in milliseconds (ms) to evaluate cardiac safety.
Observed value, change from baseline, and percent change from baseline in diastolic blood pressure (mmHg) as a measure of safety and tolerability. | Baseline through the treatment period and end of study at approximately week 16.
  Diastolic blood pressure measured in millimeters of mercury (mmHg) using standard clinical procedures at each study visit to assess safety and tolerability of ENV-294.
Observed value, change from baseline, and percent change from baseline in heart rate (beats per minute) as a measure of safety and tolerability. | Baseline through the treatment priod and end of study at approximately week 16.
  Heart rate measured in beats per minute (bpm) using standard clinical procedures at each study visit to assess safety and tolerability of ENV-294.
Observed value, change from baseline, and percent change from baseline in respiratory rate (breaths per minute) as a measure of safety and tolerability. | Baseline through the treatment period and end of study at approximately week 16
  Respiratory rate measured in breaths per minute using standard clinical procedures at each study visit to assess safety and tolerability of ENV-294.
Observed value, change from baseline, and percent change from baseline in body temperature (°F) as a measure of safety and tolerability. | Baseline through the treatment period and the end of the study at approximately week 16
  Body temperature measured in degrees Fahrenheit using standard clinical procedures at each study visit to assess safety and tolerability of ENV-294.
Change from baseline in hematocrit | Baseline through approximately 16 weeks (end of study)
  Assessment of change from baseline in hematocrit value to evaluate the safety and tolerability of ENV-294.
Change from baseline in red blood cell count | Baseline through approximately 16 weeks (end of study)
  Assessment of change from baseline in red blood cell (RBC) count to evaluate the safety and tolerability of ENV-294.
Change from baseline in white blood cell count with differential | Baseline through approximately 16 weeks (end of study)
  Assessment of change from baseline in white blood cell (WBC) count with differential to evaluate the safety and tolerability of ENV-294.
Change from baseline in platelet count | Baseline through approximately 16 weeks (end of study)
  Assessment of change from baseline in platelet count to evaluate the safety and tolerability of ENV-294.

SECONDARY OUTCOMES:
To assess the efficacy of ENV-294 in participants with asthma over a 12-week Treatment Period | Treatment period through the end of the study at approximately 16 weeks
  Number and percentage of participants experiencing a loss of asthma control (LOAC) event during the treatment period, defined according to protocol-specified criteria (e.g., exacerbation requiring systemic corticosteroids, hospitalization, or significant decline in lung function).
To assess the efficacy of ENV-294 in participants with asthma over a 12-week Treatment Period | From first treatment dose until the end of the study at approximately 16 weeks
  Time from the first dose of study drug to the first occurrence of a loss of asthma control (LOAC) event, as defined in the protocol.
To assess the efficacy of ENV-294 in participants with asthma over a 12-week Treatment Period | From baseline through the end of the study at approximately 16 weeks.
  Change from baseline in pre- and post-bronchodilator forced expiratory volume in 1 second (FEV₁), measured using standardized spirometry.
Plasma Cmax (maximum observed plasma concentration) of ENV-294 | At each scheduled PK collection time point during the 12-week treatment period
  Plasma concentrations of ENV-294 will be measured at specified time points following oral administration to determine the maximum observed concentration (Cmax).
Plasma Tmax (time to reach maximum plasma concentration) of ENV-294 | At each scheduled pharmacokinetic (PK) collection time point during the 12-week treatment period
  Time to reach maximum plasma concentration (Tmax) of ENV-294 will be determined from measured plasma concentrations following oral administration.
Plasma AUC (area under the concentration-time curve) of ENV-294 | At each scheduled pharmacokinetic (PK) collection time point during the 12-week treatment period
  Area under the plasma concentration-time curve (AUC) for ENV-294 will be calculated from measured plasma concentrations to assess overall drug exposure.

CONTACTS AND LOCATIONS:
Overall Officials: Gurpreet Ahluwalia, PhD, Study Director — Enveda Therapeutics
Locations (1):
- Velocity Clinical Research - Medford, Medford, Oregon, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared. The data include sensitive health information that cannot be fully de-identified under current privacy standards, and the sponsor does not plan to make IPD available outside the study team. Summary results and aggregate data will be shared publicly as required by regulation.